CLINICAL TRIAL: NCT02608697
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of CAT-2054 in Combination With Atorvastatin in Patients With Hypercholesterolemia
Brief Title: A Study to Assess the Safety and Efficacy of CAT-2054 in Combination With Atorvastatin in Patients With Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catabasis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAT-2054-201
Record Dates: First submitted 2015-11-11; First posted 2015-11-20 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: CAT-2054 or Placebo Dose 1 (Experimental): A run-in phase with 40 mg atorvastatin tablet administered daily for at least 28 days, followed by a 28-day blinded treatment phase with 250 mg CAT-2054 or placebo QD and open label 40 mg atorvastatin tablet administered daily.
  Interventions: Drug: CAT-2054; Drug: Placebo; Drug: Atorvastatin
- Group 2: CAT-2054 or Placebo Dose 2 (Experimental): A run-in phase with 40 mg atorvastatin tablet administered daily for at least 28 days, followed by a 28-day blinded treatment phase with 400 mg CAT-2054 or placebo QD and open label 40 mg atorvastatin tablet administered daily.
  Interventions: Drug: CAT-2054; Drug: Placebo; Drug: Atorvastatin
- Group 3: CAT-2054 or Placebo Dose 3 (Experimental): A run-in phase with 40 mg atorvastatin tablet administered daily for at least 28 days, followed by a 28-day blinded treatment phase with 250 mg CAT-2054 or placebo BID and open label 40 mg atorvastatin tablet administered daily.
  Interventions: Drug: CAT-2054; Drug: Placebo; Drug: Atorvastatin
- Group 4: CAT-2054 or Placebo Dose 4 (Experimental): A run-in phase with 40 mg atorvastatin tablet administered daily for at least 28 days, followed by a 28-day blinded treatment phase with 400 mg CAT-2054 or placebo BID and open label 40 mg atorvastatin tablet administered daily.
  Interventions: Drug: CAT-2054; Drug: Placebo; Drug: Atorvastatin

INTERVENTIONS:
Drug: CAT-2054
Drug: Placebo
Drug: Atorvastatin

SUMMARY:
The purpose of this placebo-controlled, double-blind study is to assess the effect of several doses of CAT-2054 on LDL-C in hypercholesterolemic patients on a stable dose of high-intensity statin, and to evaluate the safety and tolerability of different doses of CAT-2054 for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 74 years at Screening
* Hypercholesterolemia (LDL-C ≥ 70 mg/dL and < 190 mg/dL) plus a stable dose of statin for at least 4 weeks prior to Screening
* Satisfies one of the following:

  1. Female patients of childbearing potential must have used appropriate and highly effective contraception (a regimen which results in a failure rate of <1% per year) with their partners for 4 weeks prior to Screening, and remain compliant during the treatment phase and until 4 weeks after the last dose of investigational product
  2. Male patients must use an acceptable and highly effective contraceptive method during the treatment phase and until 4 weeks after the last dose of investigational product
* Body mass index (BMI) ≤45 kg/m2

Exclusion Criteria:

* History of any major cardiovascular event (stroke, TIA, MI, PTCI, CABG, hospitalization due to heart failure) within 6 months of Screening
* Type I diabetes mellitus or use of insulin
* Active peptic ulcer disease or a history of muscle disease or myopathy

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Percent change in LDL-C from baseline in patients with hypercholesterolemia. | 4 weeks

SECONDARY OUTCOMES:
Frequency of adverse events | 8 weeks
  Safety and tolerability will be assessed for all enrolled patients from the time the patient signs the informed consent through post-treatment follow-up. Safety parameters include physical exam, vital signs, clinical laboratory tests, ECGs and concomitant medications.
Percent change in TG, non-HDL-C, total cholesterol, HDL-C, apoB from baseline in patients with hypercholesterolemia | 4 weeks

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Muscle Shoals, Alabama
  - Huntington Park, California
  - Lomita, California
  - Los Angeles, California
  - Brooksville, Florida
  - Hialeah, Florida
  - Jupiter, Florida
  - Pembroke Pines, Florida
  - Winter Park, Florida
  - Chicago, Illinois
  - Evanston, Illinois
  - Indianapolis, Indiana
  - Kansas City, Kansas
  - Louisville, Kentucky
  - Auburn, Maine
  - Troy, Michigan
  - Las Vegas, Nevada
  - New York, New York
  - Rochester, New York
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Franklin, Ohio
  - Lyndhurst, Ohio
  - Marion, Ohio
  - Willoughby Hills, Ohio
  - Mt. Pleasant, South Carolina
  - Summerville, South Carolina
  - Houston, Texas
  - Orem, Utah
  - Richmond, Virginia
  - Olympia, Washington